CLINICAL TRIAL: NCT03842085
Title: Evaluation on Open-Labeled and Dose-Escalation Phase I Clinical Study of Safety and Pharmacokinetics of Recombinant Humanized Bispecific Monoclonal Antibody MBS301 for Injection in Treatment of HER2 Positive Recurrent or Metastatic Malignant Solid Tumor
Brief Title: Phase I Clinical Study of MBS301 in Treatment of HER2 Positive Recurrent or Metastatic Malignant Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBS301-CT01
Record Dates: First submitted 2019-02-02; First posted 2019-02-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: HER2-positive Recurrent or Metastatic Malignant Solid Tumor
Keywords: HER2-positive; solid tumor; MBS301
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBS301 (Experimental): Drug: Recombinant Humanized Bispecific Monoclonal Antibody MBS301
  Interventions: Drug: Recombinant Humanized Bispecific Monoclonal Antibody MBS301

INTERVENTIONS:
Drug: Recombinant Humanized Bispecific Monoclonal Antibody MBS301 — The patients confirming to the eligibility criteria will be assigned to the 8 dose groups based on the sequence of inclusion. MBS301 will be administered intravenousely on day 1 of each 21-day cycle for each patient.The first intravenous infusion for each patient will be last for 90 minutes.It could be changed to 60 minutes for the subsequent infusions if the drug is well tolerated.
  Other Names: MBS301

SUMMARY:
This is a phase I study evaluating the safety and pharmacokinetics of MBS301 after intravenous administration in patients with HER-2 positive recurrent or metastatic malignant solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2-positive recurrent or metastatic malignant solid tumor diagnosed by histopathology or cytology.
2. Patients with any types of malignant solid tumors who have progressed despite standard therapy or are intolerant of standard therapy, or for which no standard therapy exists.
3. Patients should have measurable lesions or immeasurable lesions (according to RECIST 1.1).
4. ECOG physical condition: 0 or 1 point.
5. Expected survival period exceeds 12 weeks.

Exclusion Criteria:

1. Absolute neutrophils count (ANC) is less than1.5×109/L and/or blood platelets less than 100 ×109/L and/or hemoglobin less than 9g/dL.
2. Total bilirubin is more than 1.5 ×ULN.
3. Patients without hepatic metastasis, ALT or AST is more than 1.5 ×ULN; Patients with hepatic metastasis, ALT or AST is more than 3 ×ULN.
4. Serum creatinine is more than 1.5 × ULN or estimated creatinine clearance <50 mL/min(according to Cockcroft-Gault).
5. International normalized ratio (INR) is more than 1.5 × ULN or activated partial thromboplastin time (APTT) is more than 1.5 × ULN.
6. Patient has prior treated with anthracyclineswhich accumulated dose is equivalent to adriamycin≥360mg/m2.
7. Patient has been experienced toxic reactions after previous anticancer therapy and has not recovered to Grade 0 or Grade 1 (except for hair loss).
8. Known a history with brain metastasis.
9. Have a history of liver disease of clinical significance.
10. Known to be human immunodeficiency virus (HIV) positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DLT of MBS301 | up to the third treatment cycle of the last subject was ended (each cycle is 21 days)
  Evaluate the safety of MBS301 and determine the dose limited toxicity (DLT) .
MTD of MBS301 | up to the third treatment cycle of the last subject was ended (each cycle is 21 days)
  Evaluate the safety of MBS301 and determine the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Investigate the pharmacokinetics profile(Cmax) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Maximum Plasma Concentration [Cmax]
Investigate the pharmacokinetics profile(AUC) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Area Under the Curve [AUC]
Investigate the pharmacokinetics profile(Tmax) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Time for Peak concentration[Tmax]
Investigate the pharmacokinetics profile(MRT) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Mean ResidenceTime[MRT]
Investigate the pharmacokinetics profile(T1/2) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Half-life[T1/2]
Investigate the pharmacokinetics profile(Vd) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Apparent volume of distribution[Vd]
Investigate the pharmacokinetics profile(CL) of MBS301 | At the end of Cycle 3 (each cycle is 21 days)
  Clearance[CL]
Evaluate the immunogenicity of MBS301 | screening, before the second/third cycle of administration, Cycle 1 day 15, at the end of Cycle 3 (each cycle is 21 days)
  Anti-drug antibody (ADA)
Evaluate the objective response rate (ORR)of MBS301 | up to approximately 2 years
  objective response rate (ORR)
Evaluate the duration of response (DoR) of MBS301 | up to approximately 2 years
  duration of response (DoR)
Evaluate the disease control rate (DCR) of MBS301 | up to approximately 2 years
  disease control rate (DCR)
Evaluate the progression free survival (PFS) of MBS301 | up to approximately 2 years
  progression free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China